CLINICAL TRIAL: NCT01370291
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for First-episode Schizophrenia Patients:A Double-blinded , Randomized and Functional Magnetic Resonance Imaging (fMRI)Study
Brief Title: Repetitive Transcranial Magnetic Stimulation for First-episode Schizophrenia Patients
Acronym: rTMSfMRI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, fengshufang, Fourth Military Medical University, Department of Psychiatry, Xi Jing hospital, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20110526-08
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Schizophrenia
Keywords: rTMS; Risperidone
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- active Risperidone and active rTMS (Active Comparator): active Risperidone and active rTMS for the first-episode schizophrenia patients
  Interventions: Other: active Risperidone and active rTMS
- active rTMS and sham Risperidone (Experimental): active rTMS and sham Risperidone for the first-episode schizophrenia
  Interventions: Other: active rTMS and sham Risperidone
- sham rTMS and active Risperidone (Sham Comparator): sham rTMS and active Risperidone for the first-episode schizophrenia patients
  Interventions: Other: sham rTMS and active Risperidone

INTERVENTIONS:
Other: active Risperidone and active rTMS — active Risperidone:------- active rTMS:auditory hallucinations:low-frequency(1Hz)applied over the left temporoparietal cortex(LTPC) negative symptoms:high-frequency（10Hz）applied over the left temporoparietal cortex(LTPC)
  Other Names: Risperidone:Xian-Janssen pharmaceutical ltd; rTMS:MagVenture
  Arms: active Risperidone and active rTMS
Other: active rTMS and sham Risperidone — active Risperidone:------- ; active rTMS:auditory hallucinations:low-frequency(1Hz)applied over the left temporoparietal cortex(LTPC); negative symptoms:high-frequency（10Hz）applied over the left temporoparietal; cortex(LTPC)
  Other Names: Risperidone:Xian-Janssen pharmaceutical ltd; rTMS: MagVenture
  Arms: active rTMS and sham Risperidone
Other: sham rTMS and active Risperidone — active Risperidone:------- ; active rTMS:auditory hallucinations:low-frequency(1Hz)applied over the left temporoparietal cortex(LTPC); negative symptoms:high-frequency（10Hz）applied over the left temporoparietal; cortex(LTPC)
  Other Names: Risperidone:Xian-Janssen pharmaceutical ltd; rTMS: MagVenture
  Arms: sham rTMS and active Risperidone

SUMMARY:
The aim of the study is to evaluate the effects of repetitive transcranial magnetic stimulation(rTMS)in the first-episode Schizophrenic patients: the clinical and MRI findings

ELIGIBILITY:
Inclusion Criteria:

* Age between 16-45 years
* Diagnosis of schizophrenia according to DSM-IV criteria(by a board-certified psychiatrist)
* PANSS>=60
* First episode, and the patients haven't use any antipsychotic drugs

Exclusion Criteria:

* Suicide risk
* Diagnose of substance abuse/dependance
* Severe uncontrolled organic disease that may interfere in the patient´s participation in the study
* Contraindication to TMS:

  1. Implanted pacemaker
  2. Medication pump
  3. Vagal stimulator
  4. Deep brain stimulator
  5. Metallic hardware in the head or scalp: shrapnel, surgical clips, or fragments from welding
  6. Signs of increased intracranial pressure
* Pregnancy or lactating; note that a negative pregnancy test will be required if the patient is a female in reproductive years
* Estimated IQ less than 80
* Have a sibling or parent with epilepsy

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
PANSS | 1-6 weeks

SECONDARY OUTCOMES:
Total AHRS score | 1-6 weeks
HAMD Score | 1-6 weeks
CGI | 1-6 weeks
fMRI | 0,6 week

CONTACTS AND LOCATIONS:
Overall Officials: Qingrong Tan, Ph.D, Study Director — Department of Psychiatry, Xi Jing hospital, Xi'an, China
Locations (1):
- Yun chun Chen, Xi'an, Shaanxi, China